CLINICAL TRIAL: NCT02874287
Title: Hydroxychloroquine Assessment of Management Study in Coronary Artery Disease After Angiography.
Brief Title: Efficacy Study of Hydroxychloroquine to Treat High-risk Coronary Artery Disease.
Acronym: CHANGAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRS-2016-011
Record Dates: First submitted 2016-08-09; First posted 2016-08-22 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Hydroxychloroquine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Other): Subjects are treated with hydroxychloroquine sulfate tablets.All the subjects are treated with guideline-based secondary prevention of coronary heart disease medications.
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets
- placebo (Other): Subjects are treated with placebo tablets. All the subjects are treated with guideline-based secondary prevention of coronary heart disease medications.
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets — Subjects are treated with oral hydroxychloroquine sulfate tablets 200mg twice daily for 20 weeks. All the interventions are built on the guideline-based secondary prevention of coronary heart disease medications.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo Tablets — Subjects are treated with oral placebo tablets 200mg twice daily for 20 weeks. All the interventions are built on the guideline-based secondary prevention of coronary heart disease medications.
  Other Names: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate whether treated with hydroxychloroquine could improve therapeutic effect for patients with high-risk coronary artery disease.

DETAILED DESCRIPTION:
This double blind, placebo, randomized controlled trial is going to assess if hydroxychloroquine could improve the high sensitivity C-reaction protein, blood lipid, blood glucose and blood pressure, also whether hydroxychloroquine could affect the secretion of inflammatory cytokines and the M1/M2 phenotype polarization of macrophages in patients with high-risk coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed coronary artery disease by coronary angiography or CT angiography.
* coronary artery disease with hypertension or diabetes or hyperlipidaemia(LDL>1.8mmol/L)
* High sensitivity C-reactive protein >1mg/L.
* On guideline-based secondary prevention of coronary heart disease medications≥1 months.
* No use of steroids, antibiotics, immunosuppressors a week before treatment.

Exclusion Criteria:

* Retinal disease.
* Chronic hepatopathy(ALT>120U/L).
* Renal dysfunction (eGFR<60).
* Moderately severe anemia, thrombocytopenia and leukocytopenia.
* Other contraindications for hydroxychloroquine.
* Active hemorrhage.
* Cancer or life expectancy< a year.
* New York Heart Association (NYHA) functional class≥class III, Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting in plan.
* Pregnancy and lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
change of fasting high sensitivity C-reactive protein | change from baseline at the 16th week, 39th week, 55th week.

SECONDARY OUTCOMES:
change of blood pressure | change from baseline at the 12th week, 20th week.
change of fasting blood lipid | change from baseline at the 12th week, 20th week.
change of fasting blood glucose | change from baseline at the 12th week, 20th week.
change of fasting insulin | change from baseline at the 12th week, 20th week.
change of echocardiogram | change from baseline at the 12th week, 20th week.
change of fasting Interleukin 6 | change from baseline at the 12th week, 20th week.
change of fasting tumor necrosis factor | change from baseline at the 12th week, 20th week.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Wu, Professor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

REFERENCES:
- [Background] Rho YH, Oeser A, Chung CP, Milne GL, Stein CM. Drugs Used in the Treatment of Rheumatoid Arthritis: Relationship between Current Use and Cardiovascular Risk Factors. Arch Drug Inf. 2009 Jun;2(2):34-40. doi: 10.1111/j.1753-5174.2009.00019.x. PMID 19684849
- [Background] Kim WU, Seo YI, Park SH, Lee WK, Lee SK, Paek SI, Cho CS, Song HH, Kim HY. Treatment with cyclosporin switching to hydroxychloroquine in patients with rheumatoid arthritis. Ann Rheum Dis. 2001 May;60(5):514-7. doi: 10.1136/ard.60.5.514. PMID 11302876
- [Background] Desai RJ, Eddings W, Liao KP, Solomon DH, Kim SC. Disease-modifying antirheumatic drug use and the risk of incident hyperlipidemia in patients with early rheumatoid arthritis: a retrospective cohort study. Arthritis Care Res (Hoboken). 2015 Apr;67(4):457-66. doi: 10.1002/acr.22483. PMID 25302481
- [Background] Achuthan S, Ahluwalia J, Shafiq N, Bhalla A, Pareek A, Chandurkar N, Malhotra S. Hydroxychloroquine's Efficacy as an Antiplatelet Agent Study in Healthy Volunteers: A Proof of Concept Study. J Cardiovasc Pharmacol Ther. 2015 Mar;20(2):174-80. doi: 10.1177/1074248414546324. Epub 2014 Aug 14. PMID 25125385
- [Background] Mercer E, Rekedal L, Garg R, Lu B, Massarotti EM, Solomon DH. Hydroxychloroquine improves insulin sensitivity in obese non-diabetic individuals. Arthritis Res Ther. 2012 Jun 7;14(3):R135. doi: 10.1186/ar3868. PMID 22676348
- [Background] Capel RA, Herring N, Kalla M, Yavari A, Mirams GR, Douglas G, Bub G, Channon K, Paterson DJ, Terrar DA, Burton RA. Hydroxychloroquine reduces heart rate by modulating the hyperpolarization-activated current If: Novel electrophysiological insights and therapeutic potential. Heart Rhythm. 2015 Oct;12(10):2186-94. doi: 10.1016/j.hrthm.2015.05.027. Epub 2015 May 27. PMID 26025323
- [Background] Ben-Chetrit E, Fischel R, Hinz B, Levy M. The effects of colchicine and hydroxychloroquine on the cyclo-oxygenases COX-1 and COX-2. Rheumatol Int. 2005 Jun;25(5):332-5. doi: 10.1007/s00296-004-0442-4. Epub 2004 Feb 13. PMID 14963695
- [Background] Wasko MC, Hubert HB, Lingala VB, Elliott JR, Luggen ME, Fries JF, Ward MM. Hydroxychloroquine and risk of diabetes in patients with rheumatoid arthritis. JAMA. 2007 Jul 11;298(2):187-93. doi: 10.1001/jama.298.2.187. PMID 17622600
- [Background] Solomon DH, Garg R, Lu B, Todd DJ, Mercer E, Norton T, Massarotti E. Effect of hydroxychloroquine on insulin sensitivity and lipid parameters in rheumatoid arthritis patients without diabetes mellitus: a randomized, blinded crossover trial. Arthritis Care Res (Hoboken). 2014 Aug;66(8):1246-51. doi: 10.1002/acr.22285. PMID 24470436
- [Background] Gottenberg JE, Ravaud P, Puechal X, Le Guern V, Sibilia J, Goeb V, Larroche C, Dubost JJ, Rist S, Saraux A, Devauchelle-Pensec V, Morel J, Hayem G, Hatron P, Perdriger A, Sene D, Zarnitsky C, Batouche D, Furlan V, Benessiano J, Perrodeau E, Seror R, Mariette X. Effects of hydroxychloroquine on symptomatic improvement in primary Sjogren syndrome: the JOQUER randomized clinical trial. JAMA. 2014 Jul 16;312(3):249-58. doi: 10.1001/jama.2014.7682. PMID 25027140
- [Background] Koch MW, Zabad R, Giuliani F, Hader W Jr, Lewkonia R, Metz L, Wee Yong V. Hydroxychloroquine reduces microglial activity and attenuates experimental autoimmune encephalomyelitis. J Neurol Sci. 2015 Nov 15;358(1-2):131-7. doi: 10.1016/j.jns.2015.08.1525. Epub 2015 Aug 28. PMID 26344560
- [Background] Hage MP, Al-Badri MR, Azar ST. A favorable effect of hydroxychloroquine on glucose and lipid metabolism beyond its anti-inflammatory role. Ther Adv Endocrinol Metab. 2014 Aug;5(4):77-85. doi: 10.1177/2042018814547204. PMID 25343023
- [Background] Al-Bari MA. Chloroquine analogues in drug discovery: new directions of uses, mechanisms of actions and toxic manifestations from malaria to multifarious diseases. J Antimicrob Chemother. 2015;70(6):1608-21. doi: 10.1093/jac/dkv018. Epub 2015 Feb 17. PMID 25693996
- [Background] Detert J, Klaus P, Listing J, Hohne-Zimmer V, Braun T, Wassenberg S, Rau R, Buttgereit F, Burmester GR. Hydroxychloroquine in patients with inflammatory and erosive osteoarthritis of the hands (OA TREAT): study protocol for a randomized controlled trial. Trials. 2014 Oct 27;15:412. doi: 10.1186/1745-6215-15-412. PMID 25348033